CLINICAL TRIAL: NCT05393258
Title: A Pilot Study of Temporally-modulated Pulsed Radiation Therapy to Reirradiate Recurrent IDH-mutant Gliomas After Prior External Beam Radiation Therapy
Brief Title: Temporally-modulated Pulsed Radiation Therapy (TMPRT) After Prior EBRT for Recurrent IDH-mutant Gliomas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202205105
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Astrocytoma; Oligodendroglioma, Adult; Glioma, Malignant
Keywords: IDH mutant glioma; astrocytoma; oligodendroglioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioma | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: temporally-modulated pulsed radiotherapy (TMPRT) (Experimental): Patients receive TMPRT daily as 10 pulses of 0.2 Gy each with a 3-minute interval between pulses (effective dose rate = 0.0667 Gy/min) to a total dose of 54 Gy at 2 Gy per day. Treatment continues for a total of 27 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: temporally-modulated pulsed radiotherapy (TMPRT)

INTERVENTIONS:
Radiation: temporally-modulated pulsed radiotherapy (TMPRT) — Intensity modulated RT (IMRT) using single or two arc therapy will be used for RT delivery.
  Other Names: pulsed low-dose-rate RT (PLRT); pulsed reduced-dose-rate RT (PRRT)

SUMMARY:
This clinical trial studies the side effects of temporally-modulated pulsed radiation therapy (TMPRT) in patients with IDH-mutant gliomas who have previously received radiation therapy to the brain. TMPRT is a radiation technique in which radiation is delivered in multiple small doses on a specific timed interval, instead of delivering one large dose at one time. This technique may improve efficacy while reducing toxicity and improving patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent IDH-mutant gliomas (either astrocytoma or oligodendroglioma) with prior external beam radiation therapy (EBRT) to the same region. The recurrent tumor may be either histologically confirmed or based on clinical assessment. Any number of prior recurrences is allowed.
* Maxium tumor diameter of 7 cm or less.
* Prior EBRT is ≥ 2 years ago.
* The region for reirradiation should have received at least 45 Gy from the prior EBRT but no more than 75 Gy. The prior EBRT could be either photon-based or proton-based.
* Prior SRS to the same region is permitted as long as the cumulative dose of EBRT plus SRS is no more than 75 Gy. The prior SRS should be completed at least 6 months ago.
* Life expectancy ≥ 12 months
* At least 18 years of age.
* Karnofsky performance status (KPS) of at least 70%.
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

* Leptomeningeal or metastatic involvement.
* Prior history of grade 3 or higher radiation necrosis that is at least possibly related to prior radiotherapy.
* Use of concurrent bevacizumab or other anti-VEGF-directed therapy during TMPRT is not allowed. If the patient is on bevacizumab, the patient needs to discontinue bevacizumab for at least 4 weeks prior to the start of TMPRT and remain stable. Other chemotherapy, immunotherapy, or target therapy can be used concurrently or adjuvantly at the discretion of treating physician.
* Medical contraindication to MRI (e.g., unsafe foreign metallic implants, incompatible pacemaker, inability to lie still for long periods, severe to end-stage kidney disease or on hemodialysis).
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute intolerable toxicities | From start of treatment through 3 months
  Intolerable toxicities are defined as grade 3 or higher central nervous system (CNS) adverse events at least possibly related to radiation as graded by the Common Terminology Criteria for Adverse Events v5.0 with the exception of grade 3 fatigue, headache, nausea, and vomiting. Any serious adverse event leading to discontinuation of TMPRT that is at least possibly related will be considered an intolerable toxicity.
Cumulative incidence of grade 3 or higher reirradiation-related central nervous system adverse events | From start of treatment through 1 year
  Adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

SECONDARY OUTCOMES:
Change in symptom burden as measured by M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT) | Assessed at approximately 3 months, 6 months, and 12 months after start of treatment
  The MDASI-BT consists of 23 symptom questions asking the patient to rate the severity of their symptoms in the last 24 hours. The range is an 11-point scale (0 to 10), with 0 being "not present" and 10 being "as bad as you can imagine". The symptom composite score is the average of the symptoms items, and the score ranges from 0 to 23 with a higher score indicating more severe symptoms. Symptom burden deterioration is defined as an increase of more than 1 point from baseline on the composite symptom scale.
Change in interference as measured by M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT) | Assessed at approximately 3 months, 6 months, and 12 months after start of treatment
  The MDASI-BT consists of 6 interference questions asking the participant to rate how their symptoms interfered with how they felt and functioned in the last 24 hours. The range is an 11-point scale (0 to 10), with 0 being "did not interfere" and 10 being "interfered completely". The interference composite score is the average of the 6 items on interferences, with a higher score indicating more interference. Interference deterioration is defined as an increase of more than 1 point from the baseline on the interference score.
Change in quality of life (QOL) as measured by self-reported QOL on the Linear Analog Scale Assessment (LASA) | Assessed at approximately 3 months, 6 months, and 12 months after start of treatment
  The LASA is a single-item questionnaire that asks the participants to rate their overall quality of life. The LASA scale runs from 0 (as bad as it can be) to 10 (as good as it can be).
Progression-free survival (PFS) | At one year after start of treatment
  PFS is defined as the time from start of treatment until time of disease progression or death from any cause. Progression will be evaluated per standard clinical care based on the Response Assessment in Neuro-Oncology (RANO) criteria for low-grade glioma (van dent Bent et al., 2011).
Overall survival (OS) | At one year after start of treatment
  OS is defined as the time from start of treatment until the date of death due to any cause.
Number of reirradiation adverse events | From start of treatment through month 12 follow-up

OTHER OUTCOMES:
Relative changes of different subtypes of myeloid cells | At baseline and week 6 of radiation therapy.
  Blood will be collected before the start of TMPRT and at week 6 of radiation therapy to assess for changes in myeloid cells.
Relative changes of different subtypes of circulating T-cells | At baseline and week 6 of radiation therapy.
  Blood will be collected before the start of TMPRT and at week 6 of radiation therapy to assess for changes in circulating T-cells.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu